CLINICAL TRIAL: NCT06272487
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Zilebesiran Used as Add-on Therapy in Adult Patients With High Cardiovascular Risk and Hypertension Not Adequately Controlled by Standard of Care Antihypertensive Medications
Brief Title: Zilebesiran as Add-on Therapy in Patients With High Cardiovascular Risk and Hypertension Not Adequately Controlled by Standard of Care Antihypertensive Medications (KARDIA-3)
Acronym: KARDIA-3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-AGT01-007
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: High Cardiovascular Risk; Hypertension
Keywords: High blood pressure; Hypertension; siRNA; Angiotensinogen; AGT; Cardiovascular disease; Chronic kidney disease; Uncontrolled hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zilebesiran (Experimental): Participants will receive zilebesiran on Day 1 of the 6-month double-blind (DB) treatment period. Participants must be on stable doses of at least 2, but not more than 4, antihypertensive medications for at least 30 days prior to screening and plan to remain on stable doses of these medications during screening and through the DB treatment period.
  Interventions: Drug: Zilebesiran
- Placebo (Placebo Comparator): Participants will receive placebo on Day 1 of the 6-month DB treatment period. Participants must be on stable doses of at least 2, but not more than 4, antihypertensive medications for at least 30 days prior to screening and plan to remain on stable doses of these medications during screening and through the DB treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zilebesiran — Zilebesiran administered by subcutaneous (SC) injection
  Other Names: ALN-AGT01
  Arms: Zilebesiran
Drug: Placebo — Placebo administered by SC injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of zilebesiran as add-on therapy in patients with high cardiovascular risk and hypertension not adequately controlled by standard of care antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

* History of cardiovascular (CV) disease, high CV risk, or estimated glomerular filtration rate (eGFR) ≥30 to <60 mL/min/1.73m^2
* Mean seated office SBP ≥140 mmHg and ≤170 mmHg
* 24-hour mean SBP ≥130 mmHg and ≤170 mmHg assessed by ABPM
* Must be on stable therapy with 2 to 4 classes of antihypertensive medications

Exclusion Criteria:

* Secondary hypertension
* Orthostatic hypotension
* Proteinuria >3 g/day
* Serum potassium >4.8 milliequivalents per liter (mEq/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline at Month 3 in Mean Seated Office Systolic Blood Pressure (SBP) | Baseline and Month 3

SECONDARY OUTCOMES:
Change from Baseline at Month 3 in 24-Hour Mean SBP Assessed by Ambulatory Blood Pressure Monitoring (ABPM) | Baseline and Month 3
Change from Baseline at Month 6 in Mean Seated Office SBP | Baseline and Month 6
Change from Baseline at Month 6 in 24-Hour Mean SBP Assessed by ABPM | Baseline and Month 6
Proportion of Patients with Mean Seated Office SBP <140 mmHg and/or Reduction ≥10 mmHg without Intensification of Antihypertensive Regimen at Month 6 | Month 6
Proportion of Patients with 24-hour Mean SBP assessed by ABPM <130 mmHg and/or Reduction ≥10 mmHg without Intensification of Antihypertensive Regimen at Month 6 | Month 6
Change from Baseline at Month 3 and Month 6 in Daytime and Nighttime Mean SBP and Diastolic Blood Pressure (DBP) assessed by ABPM | Baseline and Months 3 and 6
Change from Baseline at Month 3 and Month 6 in Mean Seated Office DBP | Baseline and Months 3 and 6
Change from Baseline at Month 3 and Month 6 in 24-hour Mean DBP Assessed by ABPM | Baseline and Months 3 and 6
Change from Baseline Over Time in Serum Angiotensinogen (AGT) | Baseline through Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (169):
- United States (121):
  - Clinical Trial Site, Alexander City, Alabama
  - Clinical Trial Site, Daphne, Alabama
  - Clinical Trial Site, Foley, Alabama
  - Clinical Trial Site, Huntsville, Alabama
  - Clinical Trial Site, Montgomery, Alabama
  - Clinical Trial Site, Gilbert, Arizona
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Sun City, Arizona
  - Clinical Trial Site, Tempe, Arizona
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Beverly Hills, California
  - Clinical Trial Site, Covina, California
  - Clinical Trial Site, Encinitas, California
  - Clinical Trial Site, Garden Grove, California
  - Clinical Trial Site, Huntington Beach, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Northridge, California
  - Clinical Trial Site, Pasadena, California
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, San Dimas, California
  - Clinical Trial Site, Santa Ana, California
  - Clinical Trial Site, Simi Valley, California
  - Clinical Trial Site, Vacaville, California
  - Clinical Trial Site, Van Nuys, California
  - Clinical Trial Site, West Hills, California
  - Clinical Trial Site, Colorado Springs, Colorado
  - Clinical Trial Site, Denver, Colorado
  - Clinical Trial Site, Hartford, Connecticut
  - Clinical Trial Site, Middlebury, Connecticut
  - Clinical Trial Site, Waterbury, Connecticut
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Clearwater, Florida
  - Clinical Trial Site, Coral Gables, Florida
  - Clinical Trial Site, Daytona Beach, Florida
  - Clinical Trial Site, Fort Myers, Florida
  - Clinical Trial Site, Hollywood, Florida
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Jensen Beach, Florida
  - Clinical Trial Site, Lake City, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, North Miami Beach, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Pembroke Pines, Florida
  - Clinical Trial Site, The Villages, Florida
  - Clinical Trial Site, Winter Haven, Florida
  - Clinical Trial Site, Acworth, Georgia
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Douglasville, Georgia
  - Clinical Trial Site, Gainesville, Georgia
  - Clinical Trial Site, Savannah, Georgia
  - Clinical Trial Site, Thomasville, Georgia
  - Clinical Trial Site, Boise, Idaho
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Elkhart, Indiana
  - Clinical Trial Site, Evansville, Indiana
  - Clinical Trial Site, Richmond, Indiana
  - Clinical Trial Site, El Dorado, Kansas
  - Clinical Trial Site, Newton, Kansas
  - Clinical Trial Site, Wichita, Kansas
  - Clinical Trial Site, Owensboro, Kentucky
  - Clinical Trial Site, Monroe, Louisiana
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Springfield, Massachusetts
  - Clinical Trial Site, Flint, Michigan
  - Clinical Trial Site, Roseville, Michigan
  - Clinical Trial Site, Ypsilanti, Michigan
  - Clinical Trial Site, Edina, Minnesota
  - Clinical Trial Site, Minneapolis, Minnesota
  - Clinical Trial Site, Columbus, Mississippi
  - Clinical Trial Site, Tupelo, Mississippi
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Kalispell, Montana
  - Clinical Trial Site, Lincoln, Nebraska
  - Clinical Trial Site, Omaha, Nebraska
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, Portsmouth, New Hampshire
  - Clinical Trial Site, Berlin, New Jersey
  - Clinical Trial Site, Albuquerque, New Mexico
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Charlotte, North Carolina
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Greensboro, North Carolina
  - Clinical Trial Site, Greenville, North Carolina
  - Clinical Trial Site, Monroe, North Carolina
  - Clinical Trial Site, Raleigh, North Carolina
  - Clinical Trial Site, Wilmington, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Marion, Ohio
  - Clinical Trial Site, Norman, Oklahoma
  - Clinical Trial Site, Oklahoma City, Oklahoma
  - Clinical Trial Site, Bethlehem, Pennsylvania
  - Clinical Trial Site, Camp Hill, Pennsylvania
  - Clinical Trial Site, Langhorne, Pennsylvania
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, East Providence, Rhode Island
  - Clinical Trial Site, Myrtle Beach, South Carolina
  - Clinical Trial Site, Rapid City, South Dakota
  - Clinical Trial Site, Chattanooga, Tennessee
  - Clinical Trial Site, Germantown, Tennessee
  - Clinical Trial Site, Knoxville, Tennessee
  - Clinical Trial Site, Memphis, Tennessee
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, Coppell, Texas
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, El Paso, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Shenandoah, Texas
  - Clinical Trial Site, Sherman, Texas
  - Clinical Trial Site, Splendora, Texas
  - Clinical Trial Site, Stephenville, Texas
  - Clinical Trial Site 1 - Tomball, Tomball, Texas
  - Clinical Trial Site 2 - Tomball, Tomball, Texas
  - Clinical Trial Site, Burlington, Vermont
  - Clinical Trial Site, Burke, Virginia
  - Clinical Trial Site, Manassas, Virginia
  - Clinical Trial Site, Norfolk, Virginia
  - Clinical Trial Site, Wauwatosa, Wisconsin
- Australia (10):
  - Clinical Trial Site, Bruce, Australian Capital Territory
  - Clinical Trial Site, Sydney, Australian Capital Territory
  - Clinical Trial Site, Brookvale, New South Wales
  - Clinical Trial Site, Concord, New South Wales
  - Clinical Trial Site, Kanwal, New South Wales
  - Clinical Trial Site, Kogarah, New South Wales
  - Clinical Trial Site, Sherwood, Queensland
  - Clinical Trial Site, Sippy Downs, Queensland
  - Clinical Trial Site, Garran
  - Clinical Trial Site, Perth
- Canada (10):
  - Clinical Trial Site, Winnipeg, Manitoba
  - Clinical Trial Site, Sarnia, Ontario
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Waterloo, Ontario
  - Clinical Trial Site, Chicoutimi, Quebec
  - Clinical Trial Site, Greenfield Park, Quebec
  - Clinical Trial Site, Montreal, Quebec
  - Clinical Trial Site, Québec, Quebec
  - Clinical Trial Site, Trois-Rivières, Quebec
  - Clinical Trial Site, Québec
- Puerto Rico (2):
  - Clinical Trial Site, Bayamón
  - Clinical Trial Site, Ponce
- Switzerland (4):
  - Clinical Trial Site, Basel
  - Clinical Trial Site, Geneva
  - Clinical Trial Site, Lausanne
  - Clinical Trial Site, Lucerne
- United Kingdom (22):
  - Clinical Trial Site, Luton, Bedfordshire
  - Clinical Trial Site, Fowey, Cornwall
  - Clinical Trial Site, Liskeard, Cornwall
  - Clinical Trial Site, Newquay, Cornwall
  - Clinical Trial Site, Torpoint, Cornwall
  - Clinical Trial Site, Chesterfield, Derbyshire
  - Clinical Trial Site, Plymouth, Devon
  - Clinical Trial Site, Bristol, Gloucestershire
  - Clinical Trial Site, Canterbury, Kent
  - Clinical Trial Site, Bellshill, Lanarkshire
  - Clinical Trial Site, Glasgow, Lanarkshire
  - Clinical Trial Site, Manchester, Lancashire
  - Clinical Trial Site, Leicester, Leicestershire
  - Clinical Trial Site, Hexham, Northumberland
  - Clinical Trial Site, Glasgow, Scotland
  - Clinical Trial Site, Carshalton, Surrey
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, Cardriff
  - Clinical Trial Site, Chorley
  - Clinical Trial Site, Liverpool
  - Clinical Trial Site, London
  - Clinical Trial Site, Pickering

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.